CLINICAL TRIAL: NCT02232672
Title: Choline PET/CT vs. MeAIB PET/CT. Better Detection of Bone and Lymph Node Metastases in Prostate Cancer Patients, PROSTAGE III
Brief Title: Choline PET/CT vs. MeAIB PET/CT in Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mike Allan Mortensen, MD, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MAM_PROSTAGE3
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Staging; PET/CT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MeAIB PET/CT (Experimental): Choline PET/CT and MeAIB PET/CT
  Interventions: Device: Choline PET/CT and MeAIB PET/CT

INTERVENTIONS:
Device: Choline PET/CT and MeAIB PET/CT — Choline PET/CT and MeAIB PET/CT

SUMMARY:
Prostate cancer is currently the leading newly diagnosed cancer in the industrialized world. Treatment of prostate cancer is highly dependent on the stage of the disease. Current methods for staging of bone metastases are known to be inaccurate. Staging of lymph nodes requires surgery associated with risk of bleeding etc. Prior studies from our department suggest that PET/CT is useful in staging of bone metastases in patients with prostate cancer. The aim of this study is to compare the usefulness of MeAIB PET/CT with current methods for the staging of bone and lymph node metastases in patients with newly diagnosed prostate cancer.

Better initial staging will result in better treatment of the individual patient. If we are able to develop a more accurate and non-invasive method of staging patients with undetected metastases on current staging will be spared of the side-effects associated with current treatment and staging- impotence, incontinence, radiation damage, bleeding, infection etc.

DETAILED DESCRIPTION:
1. Introduction. Cancer of the prostate (PCa) is currently the leading newly diagnosed cancer and the second most common cause of cancer deaths among men in the industrialized world . In Denmark alone more than 4000 men are yearly diagnosed with PCa . As PCa primarily affects elderly patients, one can assume that PCa will become one of the most important medical issues in the developed world due to the already high incidence combined with a growing population of elderly men.

   The aetiology of the disease is not well understood. In its most common form PCa evolves from the glandular tissue of the prostate. Metastatic spread will most commonly happen as lymphogenous spread to the regional lymph nodes or as haematogenous spread to the red bone marrow .

   Intended curative treatment of PCa is associated with considerable side effects, in particular incontinence, impotence and radiation damage to the surrounding tissues. Furthermore, over 30% of patients with organ-confined disease, which was treated with radical prostatectomy, will have biochemical relapse within 10 years . Relapse may be due to local recurrent disease suggesting poor surgical quality or poor initial staging with undetected metastases at the time of treatment.

   At diagnosis patients are stratified as having low, intermediary or high risk of dissieminatio according to D'Amico . Patients with intermediate or high risk of dissemination will be examined further with whole-body bone scintigraphy (WBS) and pelvic lymph node dissection (PLND).
2. Background.

   2.1. Current staging and limitations. WBS has been the examination of choice for evaluation of potential dissemination to bone. WBS utilizes 99mTc-labeled methylene diphosphonate (99mTc-MDP) that binds to the bone matrix formed by the osteoblasts. Gamma cameras detect the γ-radiation emitted by the decaying tracer thereby creating a 2-dimentional image depicting local osteoblast activity .

   Several limitations apply to the use of WBS in staging of patients with PCa. Sensitivity has reported as low as 39% in lesion-based analysis in patients with a low number of lesions . This combines with a low sensitivity due to many equivocal lesions caused by other bone pathology than metastasis.

   Sensitivity and specificity is improved by the use of single-photon emission computed tomography (SPECT), where the same tracer as with WBS is used to generate a three-dimensional image using a rotating gamma camera. This method also gives better anatomical information on the exact position of a potential metastasis.

   The examination of choice for the evaluation of potential metastases to lymph nodes is extended PLND . This procedure is done either prior to radiotherapy or during prostatectomy in patients with intermediate or high risk of dissemination. The optimal extent of the dissection is debated. The extended PLND performed at our institution includes the nodes in the obturator fossa, the nodes over the external iliac artery and vein, the nodes around the internal iliac artery and the nodes along the common iliac artery up to the crossing of the ureter. This dissection is assumed to include approximately 75% of lymph nodes known to harbor primary prostatic lymph node metastases . Extended PLND is surgically demanding with risk of lymphocele formation, infectious complications and severe bleeding due the lymph nodes' close proximity to the large vessels in the pelvis. All in all extended PLND is perhaps the best option for lymph node staging of PCa but it cannot be considered as optimal due to the above-mentioned issues.

   2.2 Positron Emission Tomography (PET). Positron Emission Tomography combined with Computerized Tomography (PET/CT) is a well-established tool in diagnosing and staging of several types of cancer . PET is an imaging technique where pairs of gamma rays emitted by positron-emitting radionuclide tracer are detected, producing a three-dimensional image of tracer concentration based on the amount of gamma rays emitted. The radioactive tracer is coupled to a biologically active molecule depending on the organ or metabolic process of interest . These images can then be fused with CT to create a combined functional and high-resolution anatomical image. Several tracers have been developed for use in cancer diagnostics and staging. As of now, PET/CT has no generally accepted role in the diagnosing or staging of PCa neither in Europe nor in the US .

   2.2.1 Choline. Choline is a precursor for phosphatidylcholine, a phospholipid that is integrated in the cell membrane making it a marker for cell membrane turnover and metabolism . 11C-Choline was first used as a PET tracer in 1997 . Since then many studies have been performed with 11C-Choline and later 18F-Choline (FCH) having approximately the same properties as 11C-Choline, but with a longer half-life (110 min vs. 20 min) making it more versatile in every-day use. A recent study from our department tested the use of FCH-PET/CT in detecting lymph node metastasis in 210 patients with PCa . The study concluded that FCH-PET/CT was not ideally suited for lymph node staging but could give additional information about bone metastasis. Several other investigators have also implied this , . A likely reason for the better detection of metastasis to the bone is that bone metastasis in an early stage is actually bone-marrow metastases rather than bone matrix metastasis and that it most likely that bone-marrow metastases proceed to bone matrix metastases. These will not be detectable by WBS (and probably not by CT and MRI either). Larger prospective series on the use of FCH-PET/CT for imaging of bone metastasis in PCa-patients have not yet been produced.

   2.2.2 MeAIB. α-(N-methyl-11C)-methylaminobutyric acid (MeAIB) is an amino acid analog that concentrates into cells only via the System A amino acid transport system, which has been shown to be highly upregulated in malignant cells making it a potential target for oncological imaging . The tracer has been developed by our local chief radiochemist and studies on biodistribution and dosimetry conclude that MeAIB is a tracer usable in humans with radiation doses lower than other used PET-tracers , . Clinical studies on the use of MeAIB-PET/CT in oncology are sparse , . The use of MeAIB-PET/CT in PCa has not been investigated. Unpublished data suggests that MeAIB could prove useful in diagnosing PCa because of a high uptake in prostatic tumors . Due to the short half-life of 11C (20 min.) an onsite cyclotron is required for performing the study, and thus this is possible in Odense.
3. Trial objective. To evaluate the diagnostic value of MeAIB-PET/CT in detecting bone and lymph node metastases in 30 patients with newly diagnosed PCa
4. Method. Patients included will have a choline-PET/CT perfomed as part of another project. In addition a MeAIB-PET/CT will be performed. The MeAIB PET/CT is performed with a single acquisition 1 hour after injection of tracer. All scans are performed in random order within three weeks and the images interpreted by a specialist in nuclear medicine and a specialist in radiology. Images are interpreted based on visual evaluation with supplementary measurements of SUV. Activity in lymph nodes will be recorded according to their location - external iliac vein, obturator fossa and internal iliac artery and vein.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, histologically verified PCa and
* Written consent and
* Planned extended lymph node dissection and
* PSA ≥ 20 ng/mL and/or
* Gleason score > 6 and/or
* cT-stage ≥ cT2c

Exclusion Criteria:

* Withdrawal of consent or
* Other active malign disease

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Metastases to bone (yes/no) Metastases to lymph nodes (yes/no) | 1 day (At the time of scan interpretation)

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospiatal, Odense, Denmark